CLINICAL TRIAL: NCT07294742
Title: First-in-Human Experience Using a Novel Balloon-shaped Large-Focal Pulsed Field Ablation Catheter in Persistent Atrial Fibrillation
Brief Title: Using a Novel Balloon-shaped Large-Focal Pulsed Field Ablation Catheter in Persistent Atrial Fibrillation
Acronym: PFApple-Per AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Hanxiong Liu, Professor, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFApple for PerAF
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; pulse field ablation; pulmonary vein isolation; posterior wall ablation; mitral isthmus; tricuspid isthmus
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ablation group (Experimental): All patients underwent PVI via point-to-point wide antral circumferential ablation (20-30 points, inter-point distance ≤10 mm) targeting 1-2 mm outside PV ostia (confirmed by angiography/3D mapping) to ensure contiguous, transmural lesions. Operators could optionally add linear ablation (LAPW, MI, CTI, endpoint: bidirectional block). For MI ablation, coronary sinus adjunctive ablation was done for residual epicardial connections if needed. PVI, LAPW isolation, and MI ablation were reassessed 20 minutes later; additional ablation was performed until durable isolation/block. Persistent AF post-ablation was treated with electrical cardioversion. Post-PFA voltage maps were generated to characterize lesions.
  Interventions: Device: a novel Balloon-shaped Large-Focal Pulsed Field Ablation Catheter

INTERVENTIONS:
Device: a novel Balloon-shaped Large-Focal Pulsed Field Ablation Catheter — All patients underwent PVI via point-to-point wide antral circumferential ablation. Operators could optionally perform linear ablation (LAPW, MI, CTI, endpoint: bidirectional block). For MI ablation, coronary sinus adjunctive ablation was done for residual epicardial connections if needed. PVI, LAPW isolation, and MI ablation were reassessed 20 minutes later; additional ablation was performed until durable isolation/block. Persistent AF post-ablation was treated with electrical cardioversion. Post-PFA voltage maps were generated to characterize lesions.

SUMMARY:
This clinical trial aims to evaluate the safety and effectiveness of pulmonary vein isolation (PVI) and linear ablation using a large-focal pulsed field ablation (PFA) catheter in patients with persistent atrial fibrillation (perAF). The study will address two primary questions:

1. Is the procedure safe, as determined by the absence of serious device- or procedure-related adverse events within 7 days post-ablation?
2. Is the catheter effective in creating durable lesions, as assessed by invasive electrophysiological remapping?

Study Design and Intervention

Eligible patients with perAF underwent PVI and linear ablation under general anesthesia using the PFApple large-focal PFA catheter. The catheter delivers a biphasic, bipolar pulsed electric field (1000V, 0.04 ms pulse duration) to create spherical ablation lesions.

Participant Follow-up Protocol

Enrolled participants will complete the following assessments:

1. Index Procedure: PVI and linear ablation with the PFApple PFA catheter.
2. Durability Assessment: Repeat invasive electrophysiological remapping at 3 months post-ablation to evaluate lesion durability.
3. Clinical Follow-up: Scheduled visits at 7 days, 30 days, 3 months, 6 months, and 12 months post-procedure. Atrial tachyarrhythmia recurrence is assessed via 12-lead electrocardiography at each visit and 24-hour or 7-day Holter monitoring at the 6- and 12-month time points.

DETAILED DESCRIPTION:
Introduction

Atrial fibrillation (AF) is the most common cardiac arrhythmia worldwide. Pulmonary vein isolation (PVI) is the established cornerstone therapy for symptomatic, drug-refractory AF. However, for persistent AF (PerAF), the efficacy of PVI alone is reduced compared to its effect in paroxysmal AF. Consequently, adjunctive ablation strategies beyond PVI are often employed in PerAF treatment.

Radiofrequency ablation remains the predominant conventional thermal technique for PerAF. However, its extensive application risks collateral tissue damage and procedure-related complications. These risks present significant challenges to achieving complete, transmural lesions, which may compromise overall ablation efficacy.

Pulsed field ablation (PFA) is an emerging non-thermal technology that induces rapid lesion formation via irreversible electroporation. This modality demonstrates high myocardial selectivity, effectively ablating cardiac tissue while sparing adjacent structures. Preclinical and clinical studies of PFA for PVI report durable lesions and an excellent safety profile, with no evidence of collateral damage. A PVI-plus-additional-ablation (PVI+) strategy is commonly used for PerAF to improve arrhythmia-free survival. However, data on the feasibility and safety of PFA for adjunctive PVI+ ablation remain limited. Whether PFA can enhance the safety and efficacy of PVI+ strategies in PerAF requires further investigation.

This first-in-human study aims to evaluate the feasibility and safety of a novel balloon-shaped, large-focal PFA catheter for PVI+ strategies in patients with PerAF.

Methods

Study Design This was a first-in-human, prospective, single-arm, single-center trial evaluating the safety and efficacy of a novel balloon-shaped, large-focal PFA catheter (PFapple™, EnChannel Medical, Guangdong, China) in patients with PerAF. The study was approved by the local Ethics Committee and conducted in accordance with the Declaration of Helsinki. All participants provided written informed consent.

Study Population Eligible patients were 18-75 years old with documented symptomatic PerAF (AF duration 7-365 days) who were refractory or intolerant to at least one Class I or III antiarrhythmic drug.

Procedural Workflow All procedures were performed under general anesthesia. Following femoral venous access, intravenous heparin was administered to maintain an activated clotting time ≥300 seconds. A decapolar catheter was positioned in the coronary sinus and a ventricular electrode in the right ventricle. Transseptal puncture was performed under fluoroscopic guidance.

An electroanatomic map of the left atrium and pulmonary veins was created using a PENTARAY® catheter and the CARTO 3 system (Biosense Webster). The PFA sheath was inserted and continuously flushed. The PFApple catheter was advanced into the left atrium and navigated to target sites.

PVI was performed in all patients using a wide antral circumferential, point-to-point technique. Typically, 20-30 ablation points were deployed along the PV antrum, maintaining an inter-point distance <10 mm to ensure lesion continuity and transmurality.

Additional ablation strategies were performed at the operator's discretion. Linear ablation targets included the left atrial posterior wall (LAPW), mitral isthmus (MI), or cavotricuspid isthmus (CTI), with bidirectional block as the endpoint. For MI ablation, if persistent epicardial connections were identified, adjunctive ablation within the coronary sinus was performed.

After a 20-minute waiting period, isolation and block were reassessed. Additional applications were delivered as needed. If AF persisted, electrical cardioversion was performed to restore sinus rhythm. Post-procedure voltage maps were generated to characterize the ablation sets.

Follow-up Post-ablation antiarrhythmic drug use was determined by the operator and typically discontinued after three months. Oral anticoagulation was maintained per guidelines. Structured follow-up occurred at 7 days and 3 months post-ablation, with lesion durability assessed via invasive remapping at 3 months. Additional visits were scheduled at 6 and 12 months. Arrhythmia recurrence was assessed using 12-lead ECGs at each visit and 24-hour or 7-day Holter monitoring at 3, 6, and 12 months.

Endpoints The primary safety endpoint was the incidence of primary adverse events (PAEs) within 7 days post-ablation. Later-occurring events (device/procedure-related death, atrio-esophageal fistula, PV stenosis) were also classified as PAEs. Persistent diaphragmatic paralysis or phrenic nerve palsy at 3 months were considered PAEs.

The primary efficacy endpoint was acute procedural success, defined as the proportion of patients achieving: 1) complete electrical isolation of all PVs, and 2) for those undergoing linear ablation, confirmed bidirectional block at all targeted sites (LAPW, MI, CTI).

Secondary efficacy endpoints included:

1. Acute PV isolation success rate.
2. Acute success rate of bidirectional block for each linear ablation site.
3. Durable success rate of bidirectional block for each linear ablation site at 3-month remapping.
4. One-year freedom from atrial tachyarrhythmia recurrence.

ELIGIBILITY:
Inclusion Criteria:

18 to 75 years with documented symptomatic PerAF (AF duration: 7 to 365 days), who were either refractory to or intolerant of at least one Class I or III antiarrhythmic drug and willing to provide informed consent.

Exclusion Criteria:

1. Paroxysmal atrial fibrillation (AF)
2. AF caused by electrolyte disorders, thyroid diseases, or reversible/non-cardiac etiologies
3. Patients undergoing retreatment after ablation for rapid atrial tachyarrhythmias
4. Patients with sustained ventricular tachycardia or ventricular fibrillation
5. Left atrial anteroposterior diameter > 55 mm
6. Pulmonary vein (PV) stenosis (>70%) or prior PV stent implantation
7. History of left atrial ablation or cardiac surgery (including left atrial appendage closure)
8. Implantation of permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardioverter-defibrillator (with or without biventricular pacing function)
9. Contraindications to anticoagulation, or history of coagulation or bleeding abnormalities
10. Severe pulmonary disease: severe pulmonary arterial hypertension or any pulmonary disease with severe dyspnea involving blood gas abnormalities
11. Any of the following cardiac surgeries, implants, or conditions:

    * Prosthetic heart valve
    * NYHA Class III or IV congestive heart failure, or left ventricular ejection fraction (LVEF) < 40%
    * Atrial septal defect or ventricular septal defect closure
    * Atrial myxoma, left atrial appendage device implantation or occlusion
12. History of any of the following within 3 months prior to the procedure:

    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention
    * Cardiac surgery (including coronary artery bypass grafting)
    * Hospitalization for heart failure
    * Pericarditis
13. History of any of the following within 3 months prior to the procedure:

    * Cerebral infarction or transient ischemic attack (TIA)
    * Documented thromboembolic events (e.g., confirmed by transesophageal echocardiography [TEE])
14. History of malignant tumor or expected life expectancy < 12 months
15. Mental disorders or history of mental illness with inability to cooperate independently
16. Lactating, pregnant, or women planning or potentially becoming pregnant
17. Acute or severe systemic infection, or significant abnormalities in liver/renal function
18. Participation in other interventional clinical trials, or ineligibility for enrollment as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint | 3 months post-ablation
  The primary safety endpoint of this pilot study was the occurrence of primary adverse events within 7 days after the index ablation procedure. Device- or procedure-related death, atrio-oesophageal fistula, and PV stenosis occurring more than 7 days post-ablation were also classified as primary adverse events. Diaphragmatic paralysis/phrenic nerve palsy were considered PAEs if symptoms persisted at the 3-month follow-up visit.
The primary efficacy endpoint | Immediately post-ablation
  The primary efficacy endpoint was the acute procedural success rate, defined as the proportion of patients who achieved all of the following: 1) complete electrical isolation of all PVs after PVI; 2) for patients undergoing additional linear ablation, bidirectional block confirmed at the targeted linear sites (LAPW, MI, or CTI).

SECONDARY OUTCOMES:
The secondary efficacy endpoints | One year post-ablation
  Including the acute success rate of individual ablation components, specifically: 1) PV isolation success rate (proportion of patients with complete isolation of all PVs); 2) success rate of bidirectional block for each linear ablation site (BOX, MI, CTI) in patients undergoing these procedures; 3) success rate of bidirectional block for each linear ablation site (BOX, MI, CTI) in patients undergoing these procedures at 3 months post-ablation remapping; and 4) the one-year rate of freedom from atrial tachyarrithmia reccurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third People's Hospital of Chengdu, Chengdu, China

IPD SHARING:
Plan to Share IPD: Yes
Those IPD are all data used in the primary results publication, as sharing them supports reproducible research and advances the understanding of large-focal PFA in persistent AF.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2-year sharing window post-publication
Access Criteria: 1. Eligible Recipients Qualified researchers with academic/institutional affiliation, who submit a feasible research proposal and agree to comply with data protection regulations.
  2. Access Process - Submit application (proposal, CV, IRB approval, signed DUA) to the corresponding author via designated email.